CLINICAL TRIAL: NCT02003885
Title: Effect of Desflurane on Left Ventricular Function in Remifentanil-based Anesthesia for Cardiac Surgery: Tissue Doppler Imaging of Mitral Valve Annular Velocity
Brief Title: Effect of Desflurane on Cardiac Function During Cardiac Surgery: Tissue Doppler Imaging of Mitral Valve Annular Velocity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KUH1160063
Record Dates: First submitted 2013-08-28; First posted 2013-12-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Valvular Heart Disease
Keywords: Desflurane, mitral annular velocity, tissue Doppler imaging
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desflurane increment (Experimental): increment of desflurane 0.5-1.5 MAC in remifentanil anesthesia for cardiac surgery
  Interventions: Drug: increment of desflurane

INTERVENTIONS:
Drug: increment of desflurane — After achieving stable hemodynamics and BIS 40-60 with desflurnae 0.5 MAC and remifentanil 0.7-1.0 mcg/kg/min (T1), data including S', E', A', EF, E, A and BIS are determined.
  After 10 min exposure to the increased desflurane dosage 1.0 MAC (T2), data are determiend. After 10 min exposure to the increased desflurane dosage 1.5 MAC (T3), data are determined.
  Reduction of BP is managed by the increment of phenylephrine infusion
  Other Names: Desflurane inhalation 0.5 MAC, 1.0 MAC and 1.5 MAC

SUMMARY:
The purpose of this study is to determine desflurane's dose-dependent effect on left ventricular (LV) function in cardiac surgery. The change of tissue Doppler imaging (TDI) of lateral mitral valve annular velocity at three different desflurane concentrations would be analyzed by using intraoperative transesophageal echocardiography (TEE) in cardiac surgery patients

DETAILED DESCRIPTION:
Tissue Doppler imaging (TDI ) of mitral annular velocity during the cardiac cycle has been introduced as a reliable method for analysis of systolic and diastolic LV ling-axix function , efficacy of diastolic TDI profile, including early early relaxation (E') and atrial contraction (A') and has been suggested to be useful in predicting the postoperative clinical outcomes and the impact of isoflurane on LV diastolic function.

Desflurane is widely used in cardiac surgery patients due to its beneficial effects , but many studies have shown that desflurane reduces myocardial contractility in a dose-dependent manner, and compromises left ventricular( LV) function We hypothesized that desflurane , even at a clinical dosage, would affects intraoperative LV systolic function in a dose-dependent manner and thus produce significant changes int the TDI profiles of mitral annular velocity.

So we planned to study the changes in TDI profiles of lateral mitral annular velocity at the clinical desflurane dosage during remifentanil based anesthesia for cardiac surgery

ELIGIBILITY:
Ages eligible for study : 20 years to 65 years Genders eligible for study : Both

Inclusion Criteria:

* Patients undergoing cardiac surgery

Exclusion Criteria:

* Low ejection fraction <50% in preoperative transthoracic echocardiography
* Atrial fibrillation
* Pacemaker
* Pericardial and infiltrative myocardial disease
* Mitral annular calcification, surgical rings, prosthetic mitral valves
* Lateral left ventricular regional wall motion abnormality
* Esophageal spasm, stricture, laceration, perforation, and diverticulum
* Diaphragmatic hernia
* History of extensive radiation to mediastinum
* Upper gastrointestinal bleeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Peak systolic mitral annular velocity (S') | after 10 min exposure to desflurane 0.5, 1.0 and 1.5 MAC
  Peak systolic mitral annular velocity (S') using tissue Doppler imaging By using pulsed Doppler with the sample volume positioned at the lateral mitral valve (MV)ring in the midesophageal 4-chamber view, S' would be determined just after the 10 min-exposure to each concentration of desflurane, 0.5 MAC, 1.0 MAC and 1.5 MAC (T1, T2 and T3, respectively)

SECONDARY OUTCOMES:
diastolic mital annular veocities (E' and A'), ejection fraction (EF), Bispectral index | after 10 min exposure to desflurane 0.5, 1.0 and1.5 MAC
  Peak mitral annular velocity during early diastole (E'): By using pulsed Doppler with the sample volume positioned at the lateral MV ring in the midesophageal 4-chamber view, Peak mitral annular velocity during atrial contraction(A'): By using pulsed Doppler with the sample volume positioned at the lateral MV ring in the midesophageal 4-chamber view, ejection fraction (EF): By using modified Simpson technique in the midesophageal 4-chamber view, bispectral index (BIS) peak velocity of mitral inflow during early relaxation (E): By using pulsed Doppler with the sample volume positioned at the IMV opening in the midesophageal 4-chamber view, peak velocity of mitral inflow during atrial contraction (A): By using pulsed Doppler with the sample volume positioned at the tip of MV opening in the midesophageal 4-chamber view,

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea